CLINICAL TRIAL: NCT00269217
Title: A Multicenter, Randomized, Double-Blind, "Factorial" Design Study to Evaluate the Lipid-Altering Efficacy and Safety of Coadministered MK0524B Tablets in Patients With Primary Hypercholesterolemia or Mixed Hyperlipidemia
Brief Title: Lipid Efficacy Study (0524B-022)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524B-022; MK0524B-022; 2005_098
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Primary Hypercholesterolemia; Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Niacin; MK-0524; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: niacin (+) laropiprant (+) simvastatin — Duration of Treatment 12 Weeks
  Other Names: MK0524B
Drug: Comparator: niacin (+) laropiprant — Duration of Treatment 12 Weeks
  Other Names: MK0524A
Drug: Comparator: simvastatin — Duration of Treatment 12 Weeks
  Other Names: MK0733

SUMMARY:
This is a 12-week clinical trial in patients with primary hypercholesterolemia or mixed hyperlipidemia, studying the effects of coadministered MK0524B on lipids. There will be 6 scheduled clinic visits, and 7 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 85 years of age with primary hypercholesterolemia or mixed hyperlipidemia
* LDL-C between 130 and 190 mg/L (Category I) and 130 and 160 mg/L (Category II) and triglycerides </= 350 mg/dL.

Exclusion Criteria:

* A condition which, in the opinion of the investigator, might pose a risk to the patient or interfere with participating in the study
* Patients with <80% compliance
* Patients with certain medical conditions
* Patients taking certain concomitant medications and/or with unstable doses of medications
* Or those with a history of CHD/CHD equivalent or diabetes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Coadministered MK0524B will be more efficacious in reducing LDL-C concentrations compared to MK0524A.

SECONDARY OUTCOMES:
Coadministered MK0524B will have a greater effect on HDL-C, TG, LDL-C, LDL-C:HDL-C, non-HDL-C, Apo B, and Apo A-I than simvastatin.
Coadministered MK0524B will have a greater effect on HDL-C, TG, LDL-C:HDL-C, non-HDL-C, Apo B, and Apo A-I than MK0524A.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Farnier M, Chen E, Johnson-Levonas AO, McCrary Sisk C, Mitchel YB. Effects of extended-release niacin/laropiprant, simvastatin, and the combination on correlations between apolipoprotein B, LDL cholesterol, and non-HDL cholesterol in patients with dyslipidemia. Vasc Health Risk Manag. 2014 May 7;10:279-90. doi: 10.2147/VHRM.S58694. eCollection 2014. PMID 24855368
- [Derived] Ballantyne C, Gleim G, Liu N, Sisk CM, Johnson-Levonas AO, Mitchel Y. Effects of coadministered extended-release niacin/laropiprant and simvastatin on lipoprotein subclasses in patients with dyslipidemia. J Clin Lipidol. 2012 May-Jun;6(3):235-43. doi: 10.1016/j.jacl.2011.11.004. Epub 2011 Dec 3. PMID 22658147
- [Derived] Bays HE, Shah A, Lin J, Sisk CM, Dong Q, Maccubbin D. Consistency of extended-release niacin/laropiprant effects on Lp(a), ApoB, non-HDL-C, Apo A1, and ApoB/ApoA1 ratio across patient subgroups. Am J Cardiovasc Drugs. 2012 Jun 1;12(3):197-206. doi: 10.2165/11631530-000000000-00000. PMID 22500948
- [Derived] Bays H, Shah A, Dong Q, McCrary Sisk C, Maccubbin D. Extended-release niacin/laropiprant lipid-altering consistency across patient subgroups. Int J Clin Pract. 2011 Apr;65(4):436-45. doi: 10.1111/j.1742-1241.2010.02620.x. PMID 21401833
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/policies-perspectives.html